CLINICAL TRIAL: NCT00727415
Title: A Prospective Multicenter Pilot Trial to Evaluate the Efficacy of a Treatment With Fludarabine, Cyclophosphamide, Lenalidomide (FCL) for Advanced Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) Patients.
Brief Title: Lenalidomide, Fludarabine & Cyclophosphamide in Advanced Chronic Lymphocytic Leukemia Not Responding to Therapy
Acronym: LLC0606
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLC0606; LLC0606 (Other: GIMEMA); 2006-006185-42 (EudraCT Number)
Record Dates: First submitted 2008-08-01; First posted 2008-08-04 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: advanced or progressive chronic lymphocytic leukemia; Lenalidomide; Fludarabine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine phosphate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cyclophosphamide — All patients will receive six monthly courses of FCL schedule consisting of three days of Fludarabine and Cyclophosphamide administration (d1-d3) combined with 14 days of Lenalidomide administration (d1-d14).
Drug: Fludarabine phosphate — All patients will receive six monthly courses of FCL schedule consisting of three days of Fludarabine and Cyclophosphamide administration (d1-d3) combined with 14 days of Lenalidomide administration (d1-d14).
Drug: Lenalidomide — All patients will receive six monthly courses of FCL schedule consisting of three days of Fludarabine and Cyclophosphamide administration (d1-d3) combined with 14 days of Lenalidomide administration (d1-d14).
  In the first phase of the study, the dose of Lenalidomide given with FC will be gradually escalated to reach the MTD. In the second phase of the study, FC will be given in combination with the Lenalidomide escalated to the MTD or the maximum planned dose.

SUMMARY:
This is a phase I - II multicenter, non-comparative, open label study in patients with previously treated CLL aimed at defining the MTD of Lenalidomide given in combination with Fludarabine, Cyclophosphamide and at evaluating the (CR) rate of FC given in combination with the MTD of Lenalidomide (FCL).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define the maximum tolerated dose (MTD) of Lenalidomide given in combination with FC.(Phase I)
* To evaluate the complete remission (CR) rate of FC given in combination with the MTD of Lenalidomide (FCL). (Phase II)

Secondary

* To define the toxicity and the infection rate of patients treated with FCL and the median number of delivered courses of FCL, overall response rate and the progression-free survival and the relationship between the response and the baseline biologic factors (IgVH, FISH, ZAP-70, CD38).
* To evaluate the overall response rate (complete and partial responses).
* To evaluate the progression-free survival.

OUTLINE: This is a phase I - II multicenter, non-comparative, open label study in patients with previously treated CLL aimed at defining the MTD of Lenalidomide given in combination with Fludarabine, Cyclophosphamide and at evaluating the (CR) rate of FC given in combination with the MTD of Lenalidomide (FCL).

All patients will receive six monthly courses of FCL schedule consisting of three days of Fludarabine and Cyclophosphamide administration (d1-d3) combined with 14 days of Lenalidomide administration (d1-d14).

After completion of study treatment, patients are followed periodically for up to 18 months.

ELIGIBILITY:
Inclusion criteria:

* Age >=18 years.
* Able to adhere to the study visit schedule and other protocol requirements.
* Patients with advanced stage or progressive CLL (NCI criteria) and relapsed or refractory disease.
* No more than 2 previous different treatment lines.
* No treatment with Campath-1H in the previous 6 months.
* Disease-free of prior malignancies for >=5 years, with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* All previous cancer therapy, including chemotherapy, immunotherapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
* ECOG performance status of <=2 at study entry.
* Laboratory test results within these ranges:

  * Serum creatinine <=1.5 mg/dL and creatinine clearance ≥60mL/min
  * Total bilirubin <=1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) <=1.5 x ULN
* Able to take low molecular weight heparin or in alternative, low- fixed-dose warfarin or, in alternative, low-dose aspirin.
* Able to understand and voluntarily sign the informed consent form.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL 10 - 14 days prior to therapy and repeated within 24 hours of starting study. FCBP must agree to use two reliable forms of contraception for at least 28 days before starting study drug; while participating in the study; and for at least 4 weeks after discontinuation from the study.
* Females must agree to abstain from breastfeeding during study participation and for at least 28 days after discontinuation from the study.
* Males must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 4 weeks following discontinuation.
* (Other details regarding pregnancy tests and contraception are reported in the chapter "Eligibility Criteria" within the study protocol).

Exclusion criteria:

* Treatment with Campath-1H during the previous 6 months.
* Concurrent use of other anti-cancer agents.
* Positive DAT with clinical and laboratory signs of hemolysis, autoimmune thrombocytopenia.
* Known positivity for HIV or active infectious hepatitis.
* Active bacterial, viral, or fungal infection requiring systemic anti-viral, antibiotic or anti-fungal therapy.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females (lactating females must agree not to breast feed while taking Lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Prior history or presence of thrombosis, thromboembolism, hearth failure or arrhythmia, neurologic disease and renal insufficiency.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum, desquamating rash while taking thalidomide or similar drugs.
* Any prior use of Lenalidomide
* Lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foa, MD, Principal Investigator — Universita Degli Studi "La Sapeinza"
Locations (23):
- Italy (23):
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Istituto di Ematologia e Oncologia Medica "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Clinica Ematologica - Università degli Studi, Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - (SA) U.O. di Oncoematologia di Nocera Inferiore-plesso ospedaliero "A. Tortora" di Pagani del DEA Nocera-Pagani, Nocera Inferiore
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Ospedale S. M. delle Croci, Ravenna
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Ospedale "Infermi", Rimini
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Universita Degli Studi "La Sapeinza", Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - U.O.C. Ematologia - Ospedale S.Eugenio, Rome
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - SS.C. di Oncoematologia - Dipartimento di Medicina Clinica e Sperimentale - Azienda Ospedaliera - S. Maria Di Terni, Terni
  - Clinica Ematologica - Policlinico Universitario, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mauro FR, Carella AM, Molica S, Paoloni F, Liberati AM, Zaja F, Belsito V, Cortellezzi A, Rizzi R, Tosi P, Spriano M, Ferretti A, Nanni M, Marinelli M, De Propris MS, Orlando SM, Vignetti M, Cuneo A, Guarini AR, Foa R. Fludarabine, cyclophosphamide and lenalidomide in patients with relapsed/refractory chronic lymphocytic leukemia. A multicenter phase I-II GIMEMA trial. Leuk Lymphoma. 2017 Jul;58(7):1640-1647. doi: 10.1080/10428194.2016.1258698. Epub 2016 Nov 23. PMID 27881039
- See also: GIMEMA Foundation Website — http://www.gimema.it

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I-II Lenalidomide: The phase I of the study, carried out at a single center (Hematology, Sapienza University of Rome) was focused at defining the MTD of lenalidomide given in combination with the FC regimen according to a 3 + 3 patient design. During the first course of treatment, lenalidomide was given to all patients at the starting dose of 2.5 mg daily (d1-d14). For the subsequent courses, the dose of lenalidomide was progressively escalated at each course, according to a 3 + 3 patient design. In 3 cohorts of 3 patients each, a daily dose of 5, 10, and 15 mg of lenalidomide was tested unless a dose limiting toxicity (DLT) was experienced.
  The presence of a persistent and severe hematologic toxicity, grade 2 tumor lysis syndrome (TLS), grade 3 tumor flare reaction (TFR), or other grade 3 toxicities was defined as DLT.
  In the second phase of the study, FC was given in combination with lenalidomide escalated from 2.5 mg to reach the MTD or the maximum planned dose of 15 mg.
Period: Phase I
Arm/Group | Phase I-II Lenalidomide
Started | 9
Completed | 7
Not Completed | 2
Not completed — Dose Limiting Toxicity | 2
Period: Phase II
Arm/Group | Phase I-II Lenalidomide
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase I-II Lenalidomide
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 66 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 40

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Lenalidomide (Phase I)
Description: Maximum tolerated dose of lenalidomide given in combination with fludarabine.
Time Frame: The MTD of Lenalinomide will be evaluated during the two courses given with the escalated dose of Lenalinomide defined by the respective dose level.
Measure: Number; unit: number of patients without DLT
Arm/Group | Phase I-II Lenalidomide
Number analyzed (Participants) | 9
number of patients without DLT
  Dose level 1 - 5 mg | 6
  Dose level 2 - 10 mg | 1

2. Primary Outcome: Overall Complete Response (CR) Rate (Phase II)
Description: Response will be assessed by clinical examination, peripheral blood, bone marrow aspirate and biopsy, radiographic evaluation. Response will be evaluated at three different levels: clinical, cytometric and molecular.
Time Frame: After 6 months from study entry (end of treatment).
Population: 7 patients coming from the phase I + 33 patients enrolled from the phase II. The whole population of phase II part of the trial is composed of a total of 40 patients.
Measure: Number; unit: percentage of patients in CR
Arm/Group | Phase I-II Lenalidomide
Number analyzed (Participants) | 40
percentage of patients in CR | 22.5

3. Secondary Outcome: Number of Patients Reaching Disease-free Survival (DSF) Overall
Description: as for outcome 2
Time Frame: After 6 months from study entry (end of treatment)
Measure: Number (95% Confidence Interval); unit: percentage of participants on DFS
Arm/Group | Phase I-II Lenalidomide
Number analyzed (Participants) | 40
percentage of participants on DFS | 35.33 [22.71 to 54.95]

4. Secondary Outcome: Toxicity as Assessed by NCI CTCAE v3.0
Description: Data from all subjects who receive any study drug will be included in the safety analyses.
Time Frame: At 24 months from study entry (end of follow-up)
Population: Fourteen (35%) patients have died.
Measure: Number; unit: Participants who died during the study
Arm/Group | Phase I-II Lenalidomide
Number analyzed (Participants) | 40
Participants who died during the study | 14

5. Secondary Outcome: Number of Patients With Severe Infections
Description: Severe infection requiring more than 2 weeks of antibiotic therapy.
Time Frame: At 24 months from study entry (end of follow-up)
Measure: Number; unit: participants with severe infecitons
Arm/Group | Phase I-II Lenalidomide
Number analyzed (Participants) | 40
participants with severe infecitons | 2

6. Secondary Outcome: Correlation Between Complete Response (CR) and Baseline Biologic Parameters (i.e., IgHV, CD38, Etc.).
Time Frame: After 6 months from study entry (end of treatment).
Measure: Number; unit: percentage of participants
Arm/Group | Phase I-II Lenalidomide
Number analyzed (Participants) | 42
percentage of participants
  CR according to IgHV mutated | 28.00
  CR according to CD19+/CD38+, <30% | 33.33
  CR according to CD19+/CD38+, >30% | 16.67
  CR according to deletion 11q and 17p, absent | 31.82

ADVERSE EVENTS:
Arm/Group | Phase I-II Lenalidomide
All-Cause Mortality (participants affected / at risk) | 14/40
Serious Adverse Events (participants affected / at risk) | 8/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I-II Lenalidomide (N=40)
Bronchopneumonia (Infections and infestations) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Multi-organi failure (General disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Intestinal obstruction (General disorders) | 1 (1)
myelodisplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No